CLINICAL TRIAL: NCT01333774
Title: Compliance With Dietary Recommendations in Obese Diabetic Patients Undergoing Acarbose Therapy
Brief Title: Influence of Different Approaches to Dietary Advising on the Effects of Acarbose Treatment in Obese Diabetic Patients Under Real-life Setting
Acronym: CATERING
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Sp. z o.o., Poland
Other Study IDs: 13928; GB0810PL (Other: Company internal)
Record Dates: First submitted 2011-04-04; First posted 2011-04-12 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Acarbose; Diet; Compliance; Advising
MeSH Terms: conditions — Diabetes Mellitus; Patient Compliance | interventions — Acarbose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Glucobay (Acarbose, BAYG5421)

INTERVENTIONS:
Drug: Glucobay (Acarbose, BAYG5421) — Patients treated with acarbose tablets under the real-life setting. Dosing regimen customised to the needs of each participating patient according to the investigators assessment

SUMMARY:
It has been recently suggested, that not the diet by itself, but also patient's adherence to dietary recommendations and all actions performed to improve dietary compliance, may be a significant factor influencing blood glucose control. There are no clinical data on the influence of different approaches to dietary advising on the effects of acarbose treatment in obese diabetic patients under real-life setting in Poland. Thus, the aim of this study was to assess the influence of different approaches to dietary advisory on the effects of acarbose treatment (reflected by changes in HbA1c) in obese DM patients. We also intended to assess the influence of different approaches to dietary advising on the appearance of potential adverse events in acarbose treated obese DM patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* age>18 years

Exclusion Criteria:

* Hypersensitivity to acarbose or any of the excipients
* age<18
* pregnancy and in nursing
* inflammatory bowel disease, colonic ulceration, partial intestinal obstruction or in patients predisposed to intestinal obstruction
* chronic intestinal diseases associated with marked disorders of digestion or absorption
* states which may deteriorate as a result of increased gas formation in the intestine, (e.g. Roemheld's syndrome [an angina pectoris-like syndrome or aggravation of an angina pectoris due to the post-prandial filling of the stomach] and larger hernias)
* hepatic and severe renal impairment (creatinine clearance <25 mL/min/ 1,73m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic diabetic patients not treated with acarbose for approx. 3 mths.
Sampling Method: Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c value between initial and final visit | approx. 3 mths after acarbose treatment initiation

SECONDARY OUTCOMES:
Number of participants with adverse events in both study groups. The influence of different approaches to dietary advising on the appearance of adverse events. | approx 3 mths after acarbose treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland